CLINICAL TRIAL: NCT05761938
Title: A Multicenter, Prospective, Real World Study of Rituximab in Frontline Therapy for Glomerulonephritis
Brief Title: A Study of Rituximab in Frontline Therapy for Glomerulonephritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Gengru Jiang, Director of Renal Division, Department of Internal Medicine, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-22-011
Record Dates: First submitted 2023-02-14; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Glomerulonephritis
Keywords: MN;MCD/FSGS;rituximab
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cohort A: pathologically confirmed membranous nephropathy
- cohort B: pathologically confirmed minimal change disease (MCD) or primary focal segmental glomerulosclerosis (FSGS)

SUMMARY:
This study included patients with glomerulonephritis who planned to receive rituximab treatment, and observed the efficacy and safety of rituximab in different glomerulonephritis in the real world. According to the pathological types of glomerulonephritis, they were divided into two cohorts : membranous nephropathy ( MN ) group or minimal change disease / focal segmental glomerulosclerosis ( MCD / FSGS ) group.

DETAILED DESCRIPTION:
A total of 100 patients with glomerulonephritis who planned to receive rituximab treatment were enrolled in the study. According to the pathological types of glomerulonephritis, they were divided into MN cohort and MCD / FSGS cohort, with 50 patients in each cohort. All eligible patients who meet the inclusion and exclusion criteria will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Primary MN, MCD/FSGS patients confirmed by biopsy
* Consistent with nephrotic syndrome ( urinary protein>3.5g/d and serum albumin< 30g/L), and the researchers consider that immunosuppressive therapy is needed
* Estimated glomerular filtration rate ( eGFR≥60 ml/min/1.73m2 )
* Patients providing written informed consent before initiation of any study-related activities

Exclusion Criteria:

* Previous treatment of rituximab
* active bacteria, fungi, tuberculosis, viral infection
* Secondary MN, MCD, FSGS ( such as active hepatitis, systemic lupus erythematosus, drugs, malignant tumors, genetic or diabetic nephropathy, etc. )
* Severe cardiac insufficiency, cardiac function in NYHA grade III above
* Severe hypertension ( blood pressure>180/110 mmHg ) that cannot be controlled by drug treatment
* Pregnant or lactating female patients
* Uncontrolled concurrent diseases, including but not limited to：

  1. HIV infected ( HIV antibody positive )
  2. HBV or HCV infection
  3. Evidence of severe or uncontrolled systemic diseases ( such as severe mental, neurological, epilepsy or dementia )
* Those currently undergoing clinical trials of other drugs
* Other patients considered unsuitable for inclusion by the researchers

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary MN, MCD/FSGS patients confirmed by biopsy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Remission Status | 12 months
  The number of subjects who achieve complete remission or partial remission in MN cohort at 12 months after treatment with Rituximab.
  CR was defined as urinary protein quantitative<0.3g and Albutein>35g/L in 24 hours.
  PR was defined as urinary protein quantitative>0.3g，but<3.5g or urinary protein decreased by 50% compared with the baseline level and the renal function was stable ( serum creatinine increased by<20% compared with the baseline level ) in 24 hours.
Remission Status | 8 weeks
  The number of subjects who achieve complete remission or partial remission in MCD/FSGS cohort at 8 weeks after treatment with Rituximab.

SECONDARY OUTCOMES:
Remission Status | 6 months
  The number of subjects who achieve complete remission or partial remission in MN cohort at 6 months after treatment with Rituximab.
Remission Status | 16 weeks
  The number of subjects who achieve complete remission or partial remission in MCD/FSGS cohort at 16 weeks after treatment with Rituximab.
Relapse | 12 months
  The number of subjects who relapse within 12 months in MCD/FSGS cohort. A relapse is defined as reappearance of Urine Protein Creatinine Ratio (based on 24-hour urine collection) > 3.5 after complete or partial remission
Incidence of adverse events (AEs) | 12 months
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: GENGRU JIANG, doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (5):
- China (5):
  - Changhai Hospital, Shanghai
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai 6th People's Hospital, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No